CLINICAL TRIAL: NCT00817492
Title: Sleep Disturbances as a Non-Traditional Risk Factor in Chronic Kidney Disease
Brief Title: Sleep Disturbances as a Non-Traditional Risk Factor in Chronic Kidney Disease- University of Illinois
Acronym: CRIC
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: #14747A; 5R01DK071696 (NIH)
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Kidney Disease
Keywords: Sleep; CKD; kidney; PSG; polysomnography; Decreased sleep time; Decreased sleep quality
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects with mild to moderate kidney disease
- 2: Healthy Control Subjects

SUMMARY:
This study will help determine the relationship between impaired sleep and chronic kidney disease, specifically to determine if sleep disturbances are a risk factor for worsening kidney function.

ELIGIBILITY:
Inclusion Criteria:

* CKD subjects will be participants in a larger study, CRIC, at the University of Illinois, Chicago
* 30 Healthy controls age and gender matched to 30 CKD subjects, regular bedtimes of at least 6h/night, sedentary lifestyle

Exclusion Criteria:

* Diabetes
* Current or previous dialysis for more than 1 month
* Uncontrolled hypertension
* Heart failure
* Liver disease
* HIV
* Hemoglobin < 10.5 g/dl
* Treatment with EProcrit, Epogen, or Aranesp
* Bone or organ transplant,
* Use of immunosuppressive drugs within past 6 months
* Current oral contraceptive use
* Current pregnancy
* Chemotherapy for malignancy within past 2 years

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Renal Clinic patients at The University of Illinois at Chicago Hospital
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2006-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | Sleep Quality was determined after PSG on all subjects were completed

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, PhD, Principal Investigator — University of Chicago; James Lash, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- The University of Illinois at Chicago, Chicago, Illinois, United States